CLINICAL TRIAL: NCT02782013
Title: Study of Progression of Hospitalized Community Acquired Pneumonia - Genetic Resistance and Susceptibility for the Evolution of Severe Sepsis
Brief Title: Study of Progression of Community Acquired Pneumonia in the Hospital
Acronym: PROGRESS
Status: Completed | Type: Observational
Sponsor: Pneumonia Research Network on Genetic Resistance and Susceptibility for the Evolution of Severe Seps (Other)
Collaborators: University of Leipzig (Other); Jena University Hospital (Other); University of Giessen (Other); University Medicine Greifswald (Other); Charite University, Berlin, Germany (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: PROGRESS-CAP
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Pneumonia; Sepsis; Shock, Septic
Keywords: community acquired pneumonia; CAP; disease progression
MeSH Terms: conditions — Pneumonia; Sepsis; Shock, Septic; Community-Acquired Pneumonia; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from EDTA whole blood, RNA from stabilized whole blood, serum, citrate plasma, stabilized EDTA plasma, urin
Oversight: Data Monitoring Committee: No

SUMMARY:
Pneumonia is a common infectious disease of the lung, often requiring treatment in the hospital. Clinical scoring systems are available, identifying patients not requiring hospitalization. However, the course of disease of patients in the hospital remains hard to predict. While most patients will recover quickly, some will, despite appropriate treatment, develop a severe course leading to sepsis and systemic responses resulting in organ dysfunction. The PROGRESS study aims to identify clinical, genetic, and other molecular markers and combinations thereof predicting a severe course of pneumonia in the hospital. Such predictors will, for instance, support decisions on earlier transfer of patients to intensive care and thus improving outcome.

DETAILED DESCRIPTION:
Pneumonia is a common infectious disease of the lung, often requiring treatment in the hospital. Clinical scoring systems are available, identifying patients not requiring hospitalization. However, the course of disease of patients in the hospital remains hard to predict. While most patients will recover quickly, some will, despite appropriate treatment, develop a severe course leading to sepsis and systemic responses resulting in organ dysfunction. The PROGRESS study aims to identify clinical, genetic and other molecular markers and combinations thereof predicting a severe course of pneumonia in the hospital. Such predictors will, for instance, support decisions on earlier transfer of patients to intensive care and thus improving outcome.

The PROGRESS study was initially approved by the ethics board of the University Hospital Jena, Friedrich-Schiller-University Jena, Germany (2403-10/08, November 6th, 2008) and subsequently by the ethics committees of all recruiting study centers.

In this observational, longitudinal case-cohort study, patients are enrolled within 48 hours of hospitalization and patient's progress is followed in much detail for up to six days thereafter. Further data are collected until discharge from the hospital. Patients are followed up on at days 28, 180, and 360 after enrollment.

Baseline assessment comprises sociodemographic, anamnestic, family history, and live style information. Upon enrollment, Pneumonia Severity Index (PSI) and CURB-65 are determined. For the day of enrollment and up to six subsequent study days routine laboratory and clinical observations and information on therapy are documented as well as data for determining the Sequential Organ Failure Assessment (SOFA) score, Systemic Inflammatory Response Syndrome (SIRS) status, and organ dysfunction. Starting with enrollment, up to six consecutive sets of biomaterials are collected comprising serum, plasma, and materials for extraction of RNA. Blood for extraction of DNA is collected once.

Follow up comprises vital status, housing situation, recurrence of pneumonia, and a quality of life questionnaire.

Analysis of cross sectional and time series data will identify clinical, genetic, and other molecular markers predicting a severe course of pneumonia in the hospital. Analysis of multilevel 'omics data in conjunction with clinical data will provide new insights into pathomechanistic details of pneumonia progression.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization with community acquired pneumonia (CAP) confirmed by pulmonary infiltrate in chest radiograph
2. Working diagnosis of CAP by enrolling physician
3. Adult patient >= 18 years of age
4. Valid informed consent form
5. At least 2 out of the five following clinical symptoms:

   * Fever
   * Cough
   * Purulent sputum
   * Shortness of breath or need for respiratory support
   * Crackling or rales on auscultation, dullness to percussion, or bronchial breathing

Exclusion Criteria:

1. Participation in this study at an earlier time
2. Hospitalization for any reason within 28 days prior to hospitalization for the current episode of CAP
3. More than 48 hours in the hospital before enrollment
4. Pregnancy
5. Breastfeeding
6. Decision on limitation of therapy before enrollment
7. Known HIV infection or AIDS
8. Anti-tumor treatment within the past six months
9. Post-stenotic pneumonia in conjunction with bronchial carcinoma
10. Therapy with corticosteroids ≥ 20mg for ≥ 14 days before enrollment
11. Non-steroidal immunosuppressive therapy within the past six months
12. Cytostatic therapy within the past six months
13. Radiation therapy within the past six months
14. Bone marrow transplant received
15. Respiratory support at home via tracheostoma
16. Cystic fibrosis
17. Active tuberculosis
18. Acute lung injury or acute respiratory distress syndrome for extrapulmonary reasons
19. Massive aspiration
20. Sepsis with extrapulmonary focus
21. Acute pulmonary embolism
22. Congestive heart failure New York Heart Association (NYHA) IV stadium
23. Liver insufficiency Child-Pugh C stadium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized for treatment of community acquired pneumonia. Patients can be enrolled in general care, intensive care, and in emergency departments.
Sampling Method: Non-Probability Sample
Enrollment: 2309 (Actual)
Dates: Start 2009-08-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Worst measure of disease severity | Between enrollment and day six
  Disease severity is operationalized by the Sequential Organ Failure Assessment (SOFA-score).

SECONDARY OUTCOMES:
All cause mortality | up to one year after enrolment
disease-specific mortality | up to one year after enrolment
duration of hospitalization | up to one year after enrolment
duration of intensive care treatment | up to one year after enrolment
duration of ventilator assisted breathing | up to one year after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Suttorp, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (64):
- Austria (2):
  - LKH-Univ. Klinikum Graz, UKIM Pulmologie, Graz
  - Allgemeines Krankenhaus der Stadt Linz, Abteilung Lungenheilkunde, Linz
- Germany (62):
  - Universitätsklinikum Aachen, Med. Klinik I (Pneumologie), Aachen
  - Evangel. Krankenhausverein, Luisenhospital, Lungenzentrum, Aachen
  - Krankenhaus Angermünde, Klinik f. Innere Medizin / Pneumologie, Angermünde
  - Krankenhaus Bad Arolsen GmbH, Innere Medizin (Herz-, Kreislauf- u. Lungendiagnostik), Bad Arolsen
  - Evangelisches Krankenhaus Bad Dürkheim, Innere Medizin, Bad Dürkheim
  - Hochtaunus-Kliniken, Medizinische Klinik III, Bad Homburg
  - Lungenklinik Ballenstedt/Harz gGmbH, Ev. Fachkrankenhaus f. Lungenkrankheiten, Ballenstedt
  - Charité - Universitätsmedizin Berlin, Zentrum Anästhesiologie und Intensivmedizin, Berlin
  - Vivantes Netzwerk f. Gesundheit GmbH Vivantes Klinikum Neukölln, Klinik f. Innere Med. - Pneumologie u.Infektiologie - Thoraxzentrum, Berlin
  - HELIOS Klinikum Berlin-Buch, Interdisziplinäres Notfallzentrum mit Rettungsstelle, Berlin
  - Evangelisches Geriatriezentrum Berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Medizinische Klinik m. S. Infektiologie und Pneumologie, Berlin
  - Humboldt-Klinikum Vivantes, Kardiologie und kons. Intensivmedizin, Berlin
  - Vivantes Klinikum Spandau, Kard., Pneum. und kons. Intensivmedizin, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe, Kardio-Pneumologie, Berlin
  - Berufsgenossenschaftl. Universitätsklinikum Bergmannsheil GmbH, Klinik f. Pneumologie, Allergologie u. Schlafmedizin, Bochum
  - Evangelische Kliniken Bonn, Betriebsstätte Johanniter Krankenhaus, Innere Medizin II, Bonn
  - Med. Klinik d. Forschungszentrum Borstel, Fachkrankenhaus f. Lungenerkrankungen, Infektionen u. Allergien, Borstel
  - Evangelisches Krankenhaus Kalk gGmbH, Innere Medizin / Pneumologie, Cologne
  - Städt. Klinikum Dessau, Innere Medizin, Dessau
  - Klinikum Dortmund gGmbH, Medizinische Klinik (Pneumologie / Infektiologie), Dortmund
  - Knappschaftskrankenhaus Dortmund, Klinik für Pneumologie, Dortmund
  - Universitätsklinikum Carl Gustav Carus, TU Dresden, Medizinische Klinik 1 - Abteilung Pneumologie, Dresden
  - SRH Wald-Klinikum Gera gGmbH, Medizinische Klinik 2, Gera
  - Uniklinikum Greifswald, Zentrum für Innere Medizin B, Greifswald
  - Krankenhaus Martha-Maria Halle-Dölau, Klinik für Innere Medizin I, Halle
  - Universitätsklinikum Halle (Saale), Klinik für Innere Medizin III (Kardiologie, Pneumologie, Intensivmedizin, Angiologie), Halle
  - Universitätsklinikum Hamburg Eppendorf, Onkologisches Zentrum, Pneumologische Studienzentrale, Hamburg
  - ASKLEPIOS Klinik Wandsbek, 1. Medizinische Abteilung, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Pneumologie, Hanover
  - Klinkum Heidenheim, Medizinische Klinik II & Innere Intensiv, Heidenheim
  - Kliniken d. Main-Taunus-Kreises, Klinik f. Pneumologie u. Allg. Innere Medizin, Hofheim
  - Universitätsklinikum des Saarlandes, Innere Medizin V, Homburg/Saar
  - Universitätsklinikum Jena, Klinik für Anästhesiologie und Intensivtherapie, Jena
  - Universitätsklinikum Jena, Zentrum für Infektionsmedizin und Krankenhaushygiene, Studienabteilung, Jena
  - St.Vincentius-Kliniken gAG, Med. Klinik IV / Pneumologie, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Medizin 1, Kiel
  - Universität Leipzig, Innere Medizin, Neurologie und Dermatologie, Pneumologie / Studiensekretariat, Leipzig
  - Klinikum St. Georg gGmbH, Klinik für Infektions-/Tropenmedizin und Nephrologie, Leipzig
  - Franziskus Krankenhaus Linz, Innere Abteilung, Linz
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Med. Klinik III (Pneumologie), Lübeck
  - St. Vincenz und Elisabeth Hospital Mainz, Innere Medizin, Mainz
  - Universitätsmedizin Mannheim, Studienkoordinierungszentrum, 1. Medizinische Klinik, Mannheim
  - Städtisches Klinikum München GmbH - Klinikum Harlaching, Klinik für Gastroent., Pneum., intern. Akut- u. Intensivmedizin, München
  - Krankenhaus München-Neuperlach, Klinik für Kardiologie, Pneumologie und Internistische Intensivmedizin, München
  - Universitätsklinikum Münster, Kardiologie 1, Münster
  - Dietrich-Bonhoeffer-Klinikum, Klinik f. Innere Medizin 2 (Abt. Pulmologie), Neubrandenburg
  - Ev. Fachkrankenhaus für Atemwegserkrankungen, Neustadt
  - Pius-Hospital Oldenburg, Klinik f. Innere Med., Abt. f. Pneumologie, Oldenburg
  - Brüderkrankenhaus St. Josef, Medizinische Klinik, Paderborn
  - Christliches Krankenhaus Quakenbrück e. V., Med. Klinik (Abtl. Pneumologie, Allergologie, Schlafmedizin), Quakenbrück
  - Universitätsklinikum Regensburg, Klinik Innere Medizin I, Intensivmedizin, Endokrinologie, Regensburg
  - Mathias-Spital Rheine, Klinik für Pneumologie und Thoraxonkologie, Rheine
  - Diakoniekrankenhaus Rotenburg(Wümme)gGmbH, Zentrum für Pneumologie, Rotenburg (Wümme)
  - Altmark-Klinikum gGmbH, Krankenhaus Salzwedel, Salzwedel
  - HELIOS Kliniken Schwerin GmbH, Klinik für Internistische und Neurologische Intensivmedizin/Stroke Unit, Schwerin
  - Krankenhaus Bethanien gGmbH Solingen, Abt. Pneumologie, Solingen
  - Kreisklinik Trostberg, Innere Abteilung, Trostberg an der Alz
  - Universitätsklinikum Ulm, Klinik für Innere Medizin II, Sudienzentrale Innere II, Sektion Pneumologie, Ulm
  - HELIOS Klinikum Wuppertal, Klinik für Intensivmedizin, Wuppertal
  - HELIOS Klinikum Wuppertal, Pneumologie, Bergisches Lungenzentrum, Wuppertal
  - Missionsärztliche Klinik GmbH Würzburg, Innere Medizin (Pneumologie), Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be made available after conclusion of the study. Participants can apply for clinical and molecular study data by sending structured project proposals to the PROGRESS board. The PROGRESS board will evaluate proposals for scientific quality, adherence to the limits set by patient's informed consent statements and by intellectual property regulations of the funding agency. Proposals shall not be denied without concrete reason.

REFERENCES:
- [Derived] Rosolowski M, Oberle V, Ahnert P, Creutz P, Witzenrath M, Kiehntopf M, Loeffler M, Suttorp N, Scholz M. Dynamics of cytokines, immune cell counts and disease severity in patients with community-acquired pneumonia - Unravelling potential causal relationships. Cytokine. 2020 Dec;136:155263. doi: 10.1016/j.cyto.2020.155263. Epub 2020 Sep 4. PMID 32896803
- [Derived] Ahnert P, Creutz P, Horn K, Schwarzenberger F, Kiehntopf M, Hossain H, Bauer M, Brunkhorst FM, Reinhart K, Volker U, Chakraborty T, Witzenrath M, Loffler M, Suttorp N, Scholz M; PROGRESS Study Group. Sequential organ failure assessment score is an excellent operationalization of disease severity of adult patients with hospitalized community acquired pneumonia - results from the prospective observational PROGRESS study. Crit Care. 2019 Apr 4;23(1):110. doi: 10.1186/s13054-019-2316-x. PMID 30947753
- [Derived] Ahnert P, Creutz P, Scholz M, Schutte H, Engel C, Hossain H, Chakraborty T, Bauer M, Kiehntopf M, Volker U, Hammerschmidt S, Loeffler M, Suttorp N; PROGRESS study group. PROGRESS - prospective observational study on hospitalized community acquired pneumonia. BMC Pulm Med. 2016 Jul 28;16(1):108. doi: 10.1186/s12890-016-0255-8. PMID 27535544
- See also: Study portal for access to electronic case report form (eCRF) — http://www.progress-cap.de/